CLINICAL TRIAL: NCT00663637
Title: Evaluation of the Safety and Efficacy of CAM (Complete Airway Management) Catheters: Phase II Study
Brief Title: Removal of Endotracheal Tube Secretions Comprehensively Until Extubation
Acronym: RESCUE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: O. M. Neotech, Inc. (Industry)
Collaborators: Saint Francis Medical Center (Unknown); Statistical Consulting (Unknown)
Responsible Party: Robert Stone RRT; Stephen Bricknell RRT, Saint Francis Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-0801
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-04

CONDITIONS: Mechanical Ventilation; Pneumonia
Keywords: endotracheal tube obstruction, occlusion; mechanical ventilation, complication; work of breathing; airway resistance; secretions; pneumonia, ventilator associated; biofilms; endotracheal tube
MeSH Terms: conditions — Pneumonia; Bites and Stings; Pneumonia, Ventilator-Associated | interventions — Complementary Therapies; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CAM (Complete Airway Management) Catheters — Prior to extubation, endotracheal tube lumen secretions are mechanically removed using CAM Rescue Cath followed by CAM Endotrach Cath.
  Other Names: CAM Rescue Cath; CAM Endotrach Cath

SUMMARY:
The purpose of this study is to measure secretion accumulation within endotracheal tubes of mechanically ventilated patients and test the efficacy, safety and clinical impact of removing the secretions using novel airway management catheters (Complete Airway Management Catheters: CAM Rescue Cath and CAM Endotrach Cath).

DETAILED DESCRIPTION:
Thirty mechanically ventilated adult patients will be managed with standard suction catheters. Just prior to extubation, their physiological parameters (including work of breathing) will be recorded and acoustic reflectometry used to measure the degree of secretion accumulation within the endotracheal tube. The endotracheal tubes will then be cleaned using the CAM Catheters (Rescue Cath followed by Endotrach Cath) and the physiological parameters and endotracheal tube reflectometry measurements repeated for comparative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving medical care in adult intensive care unit setting
* Patients who have been intubated and mechanically ventilated for at least 12 hours
* Patients intubated with an endotracheal tube with an internal diameter of 7.0 mm or greater

Exclusion Criteria:

* Patients receiving medical care in a setting not compatible with an adult intensive care unit
* Patients who have been intubated and mechanically ventilated for less than 12 hours
* Patients intubated with an endotracheal tube with an internal diameter of 6.5 mm or less
* Patients intubated with dual lumen or steel-reinforced endotracheal tubes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04

PRIMARY OUTCOMES:
work of breathing | pre-extubation

SECONDARY OUTCOMES:
endotracheal tube patency | pre-extubation

CONTACTS AND LOCATIONS:
Overall Officials: Orlando V. Morejon, MD, Study Director — Saint Francis Medical Center; Omneotech
Locations (1):
- Saint Francis Medical Center, Cape Girardeau, Missouri, United States